CLINICAL TRIAL: NCT00679237
Title: Risk Reduction in Coronary Heart Disease - a Prospective Randomized Study
Brief Title: Risk Reduction in Coronary Heart Disease
Acronym: SPREK!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Sissel Ledang, Sorlandet Hospital HF, Sorlandet Hospital HF
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-07041a (REK)
Record Dates: First submitted 2007-07-05; First posted 2008-05-16 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — Diuretics; Angiotensin-Converting Enzyme Inhibitors; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Ezetimibe; Influenza Vaccines; Metformin; glimepiride; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multifactorial intervention (Active Comparator): Smoking cessation betablocker, diuretics, ACEI, ARB, statins, ezetimibe training influenza vaccine weight reduction metformin, glimepiride, insulin
  Interventions: Behavioral: smoking cessation; Drug: betablocker, diuretics, ACEI, ARB,; Drug: statins, ezetimibe; Behavioral: training; Biological: influenza vaccine; Drug: metformin, glimepiride, insulin; Behavioral: weight reduction
- Control (No Intervention): no intervention

INTERVENTIONS:
Behavioral: smoking cessation — NRT and varenicline
  Arms: Multifactorial intervention
Drug: betablocker, diuretics, ACEI, ARB, — blood pressure control according to ESC guidelines
  Arms: Multifactorial intervention
Drug: statins, ezetimibe — Cholesterol reduction according to ESC guidelines
  Arms: Multifactorial intervention
Behavioral: training — daily walking
  Arms: Multifactorial intervention
Biological: influenza vaccine — vaccine (FLuarix, Influvac etc)
  Arms: Multifactorial intervention
Drug: metformin, glimepiride, insulin — s.glucose control according to ESC guidelines
  Arms: Multifactorial intervention
Behavioral: weight reduction — diet tips
  Arms: Multifactorial intervention

SUMMARY:
Study hypothesis: Multifactorial risk reduction in coronary heart disease can reduce the risk of new coronary heart disease and death

ELIGIBILITY:
Inclusion Criteria:

* acute myocardial infarction, CABG or PCI

Exclusion Criteria:

* Age < 18 and age > 80
* pregnant
* critical illness
* drug abuse

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
New cardiovascular events (MACE) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Serena Tonstad, dr.med., Study Chair — Ullevaal University Hospital
Locations (1):
- Sorlandet Hospital, Arendal, Norway

REFERENCES:
- [Derived] Kaldal A, Tonstad S, Jortveit J. Self-reported smoking status and exhaled carbon monoxide in secondary preventive follow-up after coronary heart events: Do our patients tell the truth? Tob Prev Cessat. 2024 Sep 25;10. doi: 10.18332/tpc/191843. eCollection 2024. PMID 39323439
- [Derived] Kaldal A, Tonstad S, Jortveit J. Sex differences in secondary preventive follow-up after coronary heart events. BMC Cardiovasc Disord. 2023 Sep 14;23(1):459. doi: 10.1186/s12872-023-03483-6. PMID 37710178
- [Derived] Kaldal A, Tonstad S, Jortveit J. Association of Troponin T measurements with long-term outcomes in patients with coronary artery disease participating in a secondary prevention trial. BMC Cardiovasc Disord. 2023 Apr 28;23(1):210. doi: 10.1186/s12872-023-03249-0. PMID 37118703
- [Derived] Kaldal A, Tonstad S, Jortveit J. Long-term hospital-based secondary prevention of coronary artery disease: a randomized controlled trial. BMC Cardiovasc Disord. 2021 Dec 16;21(1):600. doi: 10.1186/s12872-021-02426-3. PMID 34915839